CLINICAL TRIAL: NCT04982263
Title: Blood Coagulation Abnormalities in COVID-19 Patients and Correlation With Severity
Brief Title: Blood Coagulation Abnormalities in COVID-19 (Corona Virus Disease-19) Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Mohammed Abdelraheem Esmaeel, assistant professor, Sohag University
Other Study IDs: Soh-Med-21-07-34
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild cases: Patients with confirmed COVID-19 and with mild disease
  Interventions: Diagnostic Test: Blood coagulation profile
- Severe cases: Patients with confirmed COVID-19 and with severe disease
  Interventions: Diagnostic Test: Blood coagulation profile

INTERVENTIONS:
Diagnostic Test: Blood coagulation profile — Venous blood sample for measurement of blood coagulation profile

SUMMARY:
The role of the coagulation parameters in predicting the severity of COVID-19 disease will be assessed

DETAILED DESCRIPTION:
In COVID-19 patients the coagulation parameters Prothrombin concentration (PC), Activated Partial Thromboplastin Time (aPTT), D Dimer, Antithrombin III (ATIII) and Fibrinogen are measured and correlation with disease severity is to be investigated

ELIGIBILITY:
Inclusion Criteria:

● Confirmed cases with COVID 19

Exclusion Criteria:

● Known history of blood coagulopathy disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases with confirmed COVID 19 disease
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
correlation of disease severity with results of laboratory test | Baseline results of coagulation profile and baseline disease severity assessment
  The results of blood coagulation profile will be correlated with degree of severity of illness

SECONDARY OUTCOMES:
Agreement of abnormalities in coagulation profile with measured inflammatory markers | baseline measurement of inflammatory markers
  The inflammatory markers will be measured and correlation with abnormalities in coagulation profile will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Hend mohamed A Esmaeel, M.D, Principal Investigator — Sohag Univesity
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Terpos E, Ntanasis-Stathopoulos I, Elalamy I, Kastritis E, Sergentanis TN, Politou M, Psaltopoulou T, Gerotziafas G, Dimopoulos MA. Hematological findings and complications of COVID-19. Am J Hematol. 2020 Jul;95(7):834-847. doi: 10.1002/ajh.25829. Epub 2020 May 23. PMID 32282949